CLINICAL TRIAL: NCT03104543
Title: Communicating Health Information and Improving Coordination With Primary Care - an Ancillary Study of the Childhood Cancer Survivor Study
Brief Title: Communicating Health Information and Improving Coordination With Primary Care
Acronym: CHIIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); St. Jude Children's Research Hospital (Other)
Responsible Party: Principal Investigator, Eric Chow, Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 8543; R01CA204378 (NIH); P30CA015704 (NIH); RG1001538 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2018-02637 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-03-23; First posted 2017-04-07 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Hypertension; Dyslipidemias; Diabetes; Childhood Cancer
Keywords: survivor; undertreatment; adherence; self-efficacy
MeSH Terms: conditions — Hypertension; Dyslipidemias; Diabetes Mellitus; Neoplasms | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial of an educational intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): Educational materials
  Interventions: Behavioral: Education
- Test results (Active Comparator): Test results only; with delayed access to the experimental materials
  Interventions: Behavioral: Test results only

INTERVENTIONS:
Behavioral: Education — 30 minute education session; 15 minute booster session at 4 months
  Arms: Education
Behavioral: Test results only — The control group will receive a copy of test results upfront but not experimental educational materials; those will be available at 1 year
  Arms: Test results

SUMMARY:
Survivors of childhood cancer are known to be at higher risk of developing premature, serious cardiovascular disease compared with the general population. Hypertension, dyslipidemia, and diabetes increase this risk beyond that attributable to one's original cancer therapy exposures. Research has shown that childhood cancer survivors also have a high burden of underdiagnosis and undertreatment of these potentially modifiable conditions. The goal of this study is to:

1. To determine the prevalence of underdiagnosis and undertreatment of common cardiometabolic conditions (i.e., hypertension, dyslipidemia, diabetes) in survivors of childhood cancer at high-risk of future serious cardiovascular disease.
2. Among survivors who are found to be underdiagnosed or undertreated, to determine (via randomized clinical trial) the efficacy of an educational intervention to improve control of these cardiometabolic conditions.
3. Determine barriers on among survivors enrolled on the randomized trial and their primary healthcare providers that contribute to undertreatment of the study's targeted cardiometabolic conditions.

DETAILED DESCRIPTION:
What is the CHIIP Study? The CHIIP Study is for Long-Term Follow-Up (LTFU) Study participants who are more likely to experience heart problems because of their cancer treatment. We want to figure out how common high blood pressure, high blood cholesterol, and high blood sugar are among LTFU Study participants.

What will be asked of participants?

LTFU Study participants who choose to enroll in this study will be asked to:

* Answer one or two short questionnaires about their medical history, current health, mood, lifestyle, and healthcare access.
* Schedule a one-time visit for an examiner to come to their home (or another location chosen by the participant) to measure blood pressure, height, weight, waist circumference, and to draw blood to test their cholesterol and blood sugar.
* If all the test results are normal, the participant will be done with the study. If the participant has a higher than normal test result, they will remain in the study and be randomly assigned to one of two groups to learn how to improve health. A year later, participants in both groups will be asked to repeat the tests mentioned above.

What's in it for participants? Participants will have some basic health measurements done for free, including height, weight, blood pressure, and blood levels of cholesterol and sugar.

The participant and their primary care provider will receive a copy of all these test results free of cost. We hope the information we gather will provide future benefits for people who were treated for cancer as children.

ELIGIBILITY:
Inclusion Criteria:

* CCSS participant who is age ≥18 years at time of consent
* High cardiovascular risk status based on CCSS risk prediction models for cardiomyopathy and ischemic heart disease
* Able to read, write, and speak English
* Living in the U.S., within 50 miles of a designated EMSI center based on CCSS's available contact information at the time of approach.
* At least one abnormal CV condition identified on home visit: blood pressure ≥130/80 mmHg or ≥130/80 if pre-existing hypertension; LDL ≥160 mg/dL; triglyceride ≥150 mg/dL (if ≥10 hours fast) or ≥200 mg/dL (if <10 hours fast); or glucose ≥100 mg/dL if ≥8 hours fast) or ≥140 mg/dL (if <8 hours fast) or HbA1c ≥5.7% (if not known to be diabetic), HbA1c ≥7% (if known diabetic)
* Free of known self-reported ischemic heart disease or cardiomyopathy
* Have access to a telephone, computer, or smartphone to receive a phone or web video-based educational intervention

Exclusion Criteria:

* Individuals with known cardiomyopathy or ischemic heart disease based on prior CCSS surveys are excluded. While not likely to be common, participants who newly report in our study's baseline survey that they have cardiomyopathy or ischemic heart disease can have a home visit completed but will then be done with the study regardless of their home visit results.
* Not currently known to be pregnant; individuals known to be pregnant and otherwise eligible for the study can be enrolled once no longer known to be pregnant. Participants who report being pregnant AFTER randomization can remain in the study.
* Individuals receiving active cancer treatment. Participants who report starting active cancer treatment AFTER randomization can remain in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chow, MD, MPH, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
After study completion and analysis is completed, study data will join other CCSS data as a NCI-supported shared resource, available to approved external investigators.

REFERENCES:
- [Derived] Chow EJ, Chen Y, Yasui Y, Baldwin LM, Hudson MM, Muller TM, Nathan PC, Ngai SL, Ohlsen TJD, Snyder C, Syrjala KL, Tonorezos ES, Armstrong GT, Oeffinger KC. Counseling and Cardiovascular Disease Risk Factor Control in Long-Term Cancer Survivors: A Randomized Clinical Trial. JAMA Netw Open. 2026 Feb 2;9(2):e2555863. doi: 10.1001/jamanetworkopen.2025.55863. PMID 41642628
- [Derived] Chow EJ, Chen Y, Armstrong GT, Baldwin LM, Cai CR, Gibson TM, Hudson MM, McDonald A, Nathan PC, Olgin JE, Syrjala KL, Tonorezos ES, Oeffinger KC, Yasui Y. Underdiagnosis and Undertreatment of Modifiable Cardiovascular Risk Factors Among Survivors of Childhood Cancer. J Am Heart Assoc. 2022 Jun 21;11(12):e024735. doi: 10.1161/JAHA.121.024735. Epub 2022 Jun 8. PMID 35674343

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Education | Test Results
Started | 175 | 172
Completed | 126 | 138
Not Completed | 49 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education | Test Results | Total
Number analyzed (Participants) | 175 | 172 | 347
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (9.9) | 39.4 (8.9) | 40.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 93 | 182
  Male | 86 | 79 | 165
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 146 | 147 | 293
  Other race/ethnicity | 29 | 25 | 54
Undertreated hypertension [Count of Participants; unit: Participants] | 68 | 55 | 123
Undertreated dyslipidemia [Count of Participants; unit: Participants] | 79 | 80 | 159
Undertreated diabetes [Count of Participants; unit: Participants] | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Undertreatment of Hypertension (>=140/90 mmHg), Dyslipidemia (LDL >=160 mg/dL or Triglyceride >=150 mg/dL), and/or Glucose Intolerance (if Prediabetes, Hemoglobin A1c >=5.7% or Fasting Glucose >=100; if Diabetes, Hemoglobin A1c >=7%)
Description: Assess the overall probability of having any undertreated condition based on home visit measurements and blood testing
Time Frame: 1 year
Population: Analysis population includes only those with 12 month follow-up data
Measure: Number; unit: participants
Arm/Group | Education | Test Results
Number analyzed (Participants) | 126 | 138
participants
  Number of participants with undertreated hypertension at follow-up | 49 | 59
  Number of participants with undertreated dyslipidemia at follow-up | 43 | 41
  Number of participants with undertreated prediabeties / diabetes at follow-up | 48 | 54
Statistical Analysis 1: Comparison: Education vs Test Results; Test type: Superiority; p = .05, Generalized estimating equation; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.67 to 1.45]

2. Secondary Outcome: Health Knowledge
Description: Childhood cancer survivors' self-reported health knowledge (measured by questionnaire)
Time Frame: 1 year
Population: Analysis population includes only those with 12 month follow-up data
Measure: Count of Participants; unit: Participants
Arm/Group | Education | Test Results
Number analyzed (Participants) | 126 | 138
Participants
  Number participants who recalled prior anthracycline exposure correctly at follow-up | 51 | 49
  Number participants who recalled prior radiotherapy exposure correctly at follow-up | 105 | 113

3. Secondary Outcome: Self-efficacy
Description: Childhood cancer survivors' self-efficacy towards managing their healthcare (measured by questionnaire). Scale is based on work by: "Schwarzer R, Jerusalem M. Generalized Self-Efficacy scale. In: Weinman J, Wright S, Johnston M, editors. Measures in Health Psychology: A User's Portfolio. Casual and Control Beliefs. Windsor, UK:NFER-NELSON; 1995. p. 35-7." Specifically, the study used an adapted version of this scale with 5-items (4-point Likert scale) that measure perceived ability to set-goals, cope and recover from setbacks. The mean raw score for each participant was multiplied by 10 and converted to a T-score per survey developers' documentation, with 50 representing the US adult population mean, with a standard deviation of 10, and higher scores reflecting higher self-efficacy.
Time Frame: 1 year
Population: Analysis population includes only those with 12 month follow-up data
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Education | Test Results
Number analyzed (Participants) | 126 | 138
T-score | 49.5 (11.8) | 50.5 (11.3)

4. Secondary Outcome: Primary Care Provider Attitudes
Description: Healthcare providers' health knowledge and self-efficacy related to the care of childhood cancer survivors (measured by questionnaire). Specific question assesses providers' self-perceived skill in taking care of such survivors, rated from 1 (strongly disagree) to 5 (strongly agree).
Time Frame: 1 year
Population: Number of primary care providers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education | Test Results
Number analyzed (Participants) | 77 | 79
units on a scale | 3.37 (1.23) | 3.46 (1.13)
Statistical Analysis 1: Comparison: Education vs Test Results; Test type: Superiority; p = .05, t-test, 2 sided; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.47 to 0.28]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Education | Test Results
All-Cause Mortality (participants affected / at risk) | 5/175 | 0/172
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/172
Other Adverse Events (participants affected / at risk) | 0/175 | 0/172

LIMITATIONS AND CAVEATS:
New participant approaches ceased as of April 1, 2020 due to COVID-19 and inability to perform home examination visits. The study was paused until alternative study approaches were developed, with remaining subjects who had already been approached resuming baseline assessments using alternative methods starting October 2020. The final study participant had their baseline assessment completed May 2021 (n=347). Because of these delays, the study did not meet its original accrual goal (n=480).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT03104543/Prot_SAP_000.pdf